CLINICAL TRIAL: NCT00241046
Title: Letrozole in the Treatment of 1st and 2nd Line Hormone Receptor Positive Breast Cancer: Pre-therapeutic Risk Assessment
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFEM345ADE02
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Metastatic Breast Cancer
Keywords: Breast cancer; Machine learning techniques; Aromatase inhibitors; 1st line treatment; 2nd line treatment
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole

INTERVENTIONS:
Drug: Letrozole

SUMMARY:
The course of the disease in female patients with metastatic mammary carcinoma can vary greatly. In this connection, the individual prognosis depends on a complex interaction of tumor- and patient-related factors. To take account of such differences, it is necessary to employ individual methods of treatment which are suited to the course of each patient's disease. Prof. Possinger and Dr. Schmid (Charite Berlin) and Prof. Wischnewsky (University of Bremen) have developed an approach that can help to achieve this goal with the aid of computerized machine learning techniques (MLT).

The use of machine learning methods can be beneficial in oncology in two respects. On the one hand, an attempt can be made to individually estimate clinically relevant parameters like, for example, the recurrence probability or expected survival time as precisely as possible based on the established prognostic factors. And on the other hand, it may be possible with the aid of MLT to understand structural relationships between the clinical result and measured or established tumor-/patient-related variables.

To analyze the possible benefits of machine learning techniques for patients with metastatic breast cancer, the aim of study FEM-D-2 is to investigate whether it is possible to characterize those patients who either do or do not respond to a specific treatment with a precision of 90%, prospectively estimate the time until worsening of the disease under a given treatment, and classify patients in groups with favorable and poor chances of medium-term survival.

The use of inductive learning algorithms with machine learning also makes it possible to very accurately estimate the time until progression of the tumor growth. In patients who respond to letrozole therapy, the time until tumor progression depends on factors like pain, age, body mass index, disease-free interval, main localization of metastatic spread, and response to previous estrogen therapy. Only very minimal differences are found when comparing the actual time until progression of the disease and that calculated by the system (at least for survival times < 1 year). Furthermore, using machine learning techniques it has become possible to use initial data assessed before a letrozole treatment to estimate the survival time and distinguish patients with a high risk of dying soon from other patients with a more favorable prognosis.

ELIGIBILITY:
Inclusion criteria for the second-line therapy:

Patients can only take part in the study if they meet all of the following criteria:

* Histologically established mammary carcinoma
* Estrogen receptor (ER+) positive and/or progesterone receptor (PgR+) positive or ER/PgR unknown
* Postmenopausal women; defined by (at least one criterion applicable):
* Amenorrhea ≥ 5 years
* Age ≥ 60
* Age ≥ 45 with amenorrhea ≥ 12 months
* Postmenopausal LH / FSH values (according to the respective institution)
* Bilateral oophorectomy
* Patients with a primary or recurrent local advanced mammary carcinoma which cannot be curatively treated with surgical procedures or radiation therapy, or patients with a metastatic mammary carcinoma after antiestrogen pretreatment.
* Patients with a recurrence under adjuvant antiestrogen therapy (e.g. tamoxifen; with or without adjuvant chemotherapy) which was administered for at least 6 months or a recurrence within the last 12 months after adjuvant antiestrogen therapy (e.g. tamoxifen, with or without adjuvant chemotherapy) which was administered for at least 6 months or progression under palliative first-line antiestrogen therapy can be included.
* At most, a previous palliative cytostatic treatment is possible
* Measurable or assessable metastases in at least one organ system with objective proof of progression; that is, evidence of newly occurring lesions or an increase in size of preexisting lesions by more than 25% with measurable metastases or worsening with assessable changes within the last 3 months before inclusion in the study
* In the case of bone metastases, imaging methods should verify that at least one preexisting osteolysis or the lytic part of an assessable mixed lesion has increased in size, or that new measurable or assessable bone metastases have developed. In assessable mixed lesions, the measurable part must constitute at least 50% of the size of the metastasis.

If no previous images are available, the increase in bone pain in connection with the detectable, measurable osteolyses or assessable mixed metastases in the pretreatment image are regarded as progression.

* Previous radiotherapy is permitted as long as the irradiated area is not the only measurable lesion
* Estimated life expectancy of at least 12 weeks
* Performance status of 50 or higher on the Karnofsky scale or WHO grade 0-2.
* Age ≥18 years
* Written informed consent of the patient

Exclusion criteria for the second-line therapy:

Patients are not allowed to take part in the study if they meet at least one of the following criteria:

* Cerebral metastasis
* Lymphangitis carcinomatosa of the lung (> 50% of the lung affected)
* Very extensive liver metastasis (in ultrasound or CT > 33% of the liver replaced by metastases)
* Inflammatory mammary carcinoma
* Other primary malignant diseases (except in situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin)
* Patients with concomitant serious, unstable cardiac diseases (angina pectoris, arrhythmia, myocardial infarction within the last six months) or uncontrolled diabetes mellitus
* Known hypersensitivity to components of the study medication
* Exclusively osteoblastic or mixed bone metastases, with a lytic percentage < 50%, in so far as no other measurable or assessable lesions are present
* Antihormonal pretreatment with aromatase inhibitors, megestrol acetate, medroxyprogesterone, or GnRH analogues
* Treatment with a hormone replacement therapy
* Taking of non-approved substances within the past 30 days and concomitant treatment with non-approved drugs

Patients with the following pretreatments should not be included in the study (selection):

* Previous endocrine treatment of a metastatic mammary carcinoma
* Patients with adjuvant or neoadjuvant endocrine treatment with or without chemotherapy within the past 12 months
* Patients with adjuvant or neo-adjuvant endocrine antiestrogen treatment for whom a recurrence occurred during or within 12 months after the end of treatment
* Patients who received more than one regimen of a systemic chemotherapy against their advanced breast cancer

Other protocol-related inclusion / exclusion criteria may apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2002-04; Primary Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Comparison of the the individual pretherapeutic predictions from the computer or doctor with the patient data obtained in a first- or second-line treatment of metastatic breast cancer after progression of the disease

SECONDARY OUTCOMES:
Determination of the individual response at 3 monthly assessments

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis